CLINICAL TRIAL: NCT07314138
Title: MICRA-HYBRID Trial: A Randomized Controlled Trial of 'Multivessel Minimally Invasive Coronary Bypass Grafting as HYBRID Revascularization Versus Conventional Off-Pump Coronary Artery Bypass Grafting'
Brief Title: Multivessel Minimally Invasive Coronary Bypass Grafting as HYBRID Revascularization Versus Conventional Off-pump Coronary Artery Bypass Grafting
Acronym: MICRA-HYBRID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, Ferdi Akca, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL-010448
Record Dates: First submitted 2025-12-03; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease (CAD); Bypass, Cardiopulmonary; Minimally Invasive Coronary Revascularization Surgery; Off-pump Coronary Artery Bypass
Keywords: minimally invasive coronary surgery; percutaneous coronary intervention; off-pump coronary artery bypass grafting; hybrid coronary revascularization; heart surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Dual center, superiority, randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multivessel hybrid coronary revascularization (HCR) (Active Comparator): Minimally invasive coronary artery bypass surgery to the left sided coronary vessels combined with percutaneous coronary intervention to the right coronary artery.
  Interventions: Procedure: Multivessel Hybrid Coronary Revascularization
- Off-pump coronary artery bypass grafting (OPCAB) (Active Comparator): Total arterial, anaortic off-pump ccoronary artery bypass grafting through median sternotomy.
  Interventions: Procedure: Off-pump coronary arterial bypass grafting (OPCAB)

INTERVENTIONS:
Procedure: Multivessel Hybrid Coronary Revascularization — Multivessel-HCR consists of MICS revascularization of the left sided coronary vessels (LAD , Cx) combined with PCI for the RCA during the same admission or within 4 weeks postoperatively. Surgical revascularization is performed through MICS which consists of either robotically or non-robotically assisted thoracoscopic IMA harvesting followed by total arterial off-pump anastomosis of the grafts through a left anterior 3-5 cm mini-thoracotomy. PCI will be performed via radial or femoral access according to local routine and is restricted to the RCA.
  Arms: Multivessel hybrid coronary revascularization (HCR)
Procedure: Off-pump coronary arterial bypass grafting (OPCAB) — OPCAB will be performed as per clinical routine at each center through a median sternotomy. IMA harvesting (pedicled or skeletonised) follows each center's routine. An anaortic, total arterial strategy with a LIMA-LAD graft and complete revascularisation is obliged.
  Arms: Off-pump coronary artery bypass grafting (OPCAB)

SUMMARY:
The MICRA-HYBRID trial is a prospective, multicenter, randomized controlled study comparing multivessel hybrid coronary revascularization (HCR) as minimally invasive arterial bypass grafting to left-sided coronary targets (LAD and LCx) plus PCI of the RCA versus conventional off-pump coronary artery bypass grafting (OPCAB) via median sternotomy in patients with three-vessel coronary artery disease. The primary goal is to evaluate whether multivessel-HCR provides superior 30-day "textbook" clinical outcomes (mortality, MI, stroke, re-exploration for bleeding, and other complications) while improving perioperative recovery and long-term cardiovascular outcomes.

DETAILED DESCRIPTION:
Coronary artery disease remains the leading cause of cardiovascular mortality worldwide. For complex, multivessel disease, surgical revascularization via CABG or OPCAB remains the guideline-recommended standard due to superior long-term outcomes compared with PCI alone. However, traditional sternotomy CABG/OPCAB is associated with significant surgical trauma, prolonged recovery, and elevated perioperative morbidity.

Minimally invasive coronary surgery (MICS) with off-pump arterial grafting through a small thoracotomy has shown favorable short-term recovery and lower morbidity in both single and multivessel disease cases. Traditionally, MICS has been limited to grafting the left anterior descending artery (LAD), with other coronary lesions treated by PCI, known as hybrid coronary revascularization (HCR). While most studies have focused on single-vessel HCR (typically LAD), the potential long-term benefits of including the circumflex (Cx) artery in a multivessel-HCR strategy remain unexplored. Given that three-vessel CAD is the most common indication for CABG, evaluating a multivessel-HCR approach (LAD + Cx via MICS, RCA via PCI) is essential.

The MICRA-HYBRID trial will randomize 250 patients with three-vessel coronary disease eligible for complete revascularization to either multivessel-HCR or conventional total-arterial OPCAB (median sternotomy, anaortic, off-pump). The primary efficacy endpoint is a composite "Textbook Outcome" at 30 days, defined by absence of death, MI, stroke, re-exploration for bleeding, and other major complications. Secondary endpoints include individual components of the Textbook Outcome, perioperative recovery parameters (ICU/hospital length of stay, ventilator time, transfusion requirement), health-related quality of life (EQ-5D), pulmonary recovery metrics, angina class (CCS), and long-term outcomes including MACCE and target-vessel revascularization up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with three-vessel disease (either angiographic stenoses >70% or a fractional flow reserve value ≤0.80)
* Left main diameter stenosis ≥50% or a left main intravascular ultrasound minimal luminal area of ≤4.5 mm2 or fractional flow reserve value ≤0.80 combined with significant CAD of the right coronary artery

Exclusion Criteria:

A potential participant who meets any of the following criteria will be excluded from participation in this study:

* Age < 18 or > 85 years
* Chronic total occlusion of the RCA
* In-stent RCA restenosis
* RCA stenosis with high-risk clinical features requiring urgent PCI or surgical revasculari-zation.
* Reverse hybrid coronary revascularization, defined as PCI-RCA followed by surgical re-vascularization.
* Acute cardiac ischemia necessitating immediate intervention.
* EF < 30 %
* eGFR < 30 ml/min
* Indication for concomitant cardiac surgery (e.g. valve or arrhythmia surgery) or non-cardiac surgery
* Previous thoracic or cardiac surgery, mediastinal irradiation, significant trauma to the chest
* Preoperative severe end-organ dysfunction (dialysis, liver failure, respiratory failure) or cancer.
* Hemodynamically significant left subclavian stenosis
* Severe chest wall deformities
* History of pericarditis
* Body mass index > 40 Kg/m2.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Composite Absence of Adverse Events within 30 Days Postoperatively (Textbook Outcome) | 30 days postoperatively
  The primary endpoint is defined as the "Textbook Outcome," which is the composite absence, within 30 days postoperatively, of the following events:
  * Mortality
  * Re-exploration for bleeding
  * Postoperative ischemia (requiring bypass grafting or acute PCI)
  * Postoperative myocardial infarction (type 5 MI according to the fourth universal definition of myocardial infarction)
  * Cardiac tamponade (requiring surgical or percutaneous intervention)
  * Cerebrovascular accident / transient ischemic attack
  * Wound infection requiring antibiotics or intervention
  * New-onset atrial fibrillation requiring medical anti-thrombotic therapy
  * Pneumonia requiring IV or oral antibiotics
  * Placement of additional chest drains
  * Prolonged hospital stay (> 7 days) after surgery

SECONDARY OUTCOMES:
Conversion to Sternotomy | Peri-operatively
  Rate of conversion to sternotomy for minimally invasive coronary surgery (MICS) patients.
Conversion to Cardiopulmonary Bypass | Peri-operatively
  Incidence of hemodynamic support with cardiopulmonary bypass during the surgical procedures.
Intensive Care Unit (ICU) Stay | 30 days postoperatively
  Duration of ICU stay following the surgical procedure (in days).
Postoperative Hospital Stay | 30 days postoperatively
  Total length of postoperative hospital stay (in days).
Mechanical Ventilation Time | 30 days postoperatively
  Total ventilation time during the postoperative period (in hours).
Postoperative Blood Loss | 30 days postoperatively
  Total volume of postoperative blood loss (in milliliters) postoperatively.
Transfusion Requirement | 30 days postoperatively
  Need for transfusion of blood products (packed units of thrombocyt, red blood cells and plasma) during the postoperative period
Phrenic Nerve Injury | 30 days postoperatively
  Incidence of phrenic nerve injury leading to diaphragm paralysis.
Postoperative Peak Expiratory Flow (PEF) | 30 days postoperatively
  PEF measurement at Day 1 and Day 3 postoperatively, and at 4 weeks post-discharge.
Quality of Life Assessment (EQ-5D) | 1 year
  Quality of life assessment using the European Quality of Life-5 Dimensions (EQ-5D) questionnaire at baseline (screening), 2 weeks and 4 weeks postoperatively and at 12 months follow-up
Angina Assessment (CCS Classification) | 1 year
  Assessment of angina using the Canadian Cardiovascular Society (CCS) classification at baseline, discharge and every 3 months for up to 1 year
Short-term Healthcare Costs | 30 days
  Healthcare costs associated with hospitalization within 30 days postoperatively (in euros), including expenses for surgical and percutaneous procedures, diagnostic tests, ICU care, nursing days, reinterventions, complications, and post-discharge admissions (e.g., emergency visits, re-admissions, primary care consultations).
Long-term Healthcare Costs | 1 year
  Healthcare costs within 1 year postoperatively (in euros), including expenses for diagnostic tests, reinterventions, emergency visits, re-admissions, primary care consultations, repeat visits, telephone, video, and written consultations, as well as after-hours urgent care (e.g., on-call GP visits).
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 5 years
  Incidence of MACCE including mortality, stroke and myocardial infarction up to 5 years post-procedure.
Target Vessel Revascularization (TVR) | 5 year
  Incidence TVR up to 5 years post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdi Akca, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Wouter Oosterlinck, Prof. Dr. MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Pim Tonino, Prof. Dr. MD, PhD, Study Chair — Catharina Ziekenhuis Eindhoven
Locations (2):
- University Hospitals Leuven, Leuven, Vlaams Brabant, Belgium
- Catharina Hospital Eindhoven, Eindhoven, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be made available upon request to the Principal Investigator after the study's completion.

REFERENCES:
- [Background] van Steenbergen GJ, Schulz DN, Slingerland SR, Tonino PA, Soliman-Hamad MA, Dekker L, van Veghel D. Introduction of a New Method to Monitor Patient-Relevant Outcomes and Costs: Using a Quality Improvement Project in Transcatheter Aortic Valve Implantation Care as an Example. Qual Manag Health Care. 2023 Oct-Dec 01;32(4):247-256. doi: 10.1097/QMH.0000000000000401. Epub 2023 Mar 16. PMID 36940366
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for Universal Definition of Myocardial Infarction; Authors/Task Force Members Chairpersons; Thygesen K, Alpert JS, White HD; Biomarker Subcommittee; Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA; ECG Subcommittee; Chaitman BR, Clemmensen PM, Johanson P, Hod H; Imaging Subcommittee; Underwood R, Bax JJ, Bonow JJ, Pinto F, Gibbons RJ; Classification Subcommittee; Fox KA, Atar D, Newby LK, Galvani M, Hamm CW; Intervention Subcommittee; Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J; Trials & Registries Subcommittee; Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML; Trials & Registries Subcommittee; Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G; Trials & Registries Subcommittee; Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D; Trials & Registries Subcommittee; Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG); Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S; Document Reviewers; Morais J, Aguiar C, Almahmeed W, Arnar DO, Barili F, Bloch KD, Bolger AF, Botker HE, Bozkurt B, Bugiardini R, Cannon C, de Lemos J, Eberli FR, Escobar E, Hlatky M, James S, Kern KB, Moliterno DJ, Mueller C, Neskovic AN, Pieske BM, Schulman SP, Storey RF, Taubert KA, Vranckx P, Wagner DR. Third universal definition of myocardial infarction. J Am Coll Cardiol. 2012 Oct 16;60(16):1581-98. doi: 10.1016/j.jacc.2012.08.001. Epub 2012 Sep 5. No abstract available. PMID 22958960
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Modrau IS, Nielsen PH, Nielsen DV, Christiansen EH, Hoffmann T, Parner ET, Benhassen LL. Outcome of hybrid compared to conventional revascularization in multivessel coronary artery disease. Scand Cardiovasc J. 2020 Dec;54(6):376-382. doi: 10.1080/14017431.2020.1821910. Epub 2020 Sep 30. PMID 32998590
- [Background] Halkos ME, Ford L, Peterson D, Bluestein SM, Liberman HA, Kilgo P, Puskas JD, Guyton RA, Chowdhury R. The impact of hybrid coronary revascularization on hospital costs and reimbursements. Ann Thorac Surg. 2014 May;97(5):1610-5; discussion 1615-6. doi: 10.1016/j.athoracsur.2014.01.047. Epub 2014 Mar 15. PMID 24636706
- [Background] Gianoli M, de Jong AR, van der Harst P, van der Kaaij NP, Jacob KA, Suyker WJL. Cost Analysis of Robot-Assisted Versus On-Pump and Off-Pump Coronary Artery Bypass Grafting: A Single-Center Surgical and 30-Day Outcomes Comparison. Innovations (Phila). 2024 Jul-Aug;19(4):416-424. doi: 10.1177/15569845241269312. Epub 2024 Sep 12. PMID 39267423
- [Background] Michael Porter, Thomas Lee. The Strategy That Will Fix Healthcare. The Magazine.
- [Background] Zhang S, Li P, Li G, Yan Y, Sun T, Lin J, Zhang C, Liu S, Qu Z, You B. Generalized hybrid coronary revascularization vs. conventional off-pump coronary artery bypass grafting for multivessel coronary artery disease. Front Cardiovasc Med. 2025 Feb 21;12:1459072. doi: 10.3389/fcvm.2025.1459072. eCollection 2025. PMID 40060966
- [Background] Harskamp RE, Vassiliades TA, Mehta RH, de Winter RJ, Lopes RD, Xian Y, Peterson ED, Puskas JD, Halkos ME. Comparative Effectiveness of Hybrid Coronary Revascularization vs Coronary Artery Bypass Grafting. J Am Coll Surg. 2015 Aug;221(2):326-34.e1. doi: 10.1016/j.jamcollsurg.2015.03.012. Epub 2015 Mar 20. PMID 25899734
- [Background] Patel PM, Arrington RL, Jonsson A, Wei JW, Binongo J, Devireddy C, Nicholson W, Jaber W, Rinfret S, Halkos ME. Advancing the Treatment Paradigm for Multivessel Coronary Artery Disease: Hybrid Coronary Revascularization. Innovations (Phila). 2025 Jan-Feb;20(1):57-64. doi: 10.1177/15569845241311292. Epub 2025 Feb 2. PMID 39894999
- [Background] Qu W, Wei J, Binongo JN, et al. Ischemic Heart Disease HYBRID CORONARY REVASCULARIZATION PROVIDES COMPARABLE LONG-TERM OUTCOMES TO CORONARY ARTERY BYPASS GRAFTING FOR PATIENTS WITH TWO-VESSEL CORONARY DISEASE. Vol 83.; 2024.
- [Background] Xia Y, Katz AN, Forest SJ, Pyo RT, Greenberg MA, DeRose JJ Jr. Hybrid Coronary Revascularization has Improved Short-term Outcomes but Worse Mid-term Reintervention Rates Compared to CABG: A Propensity Matched Analysis. Innovations (Phila). 2017 May/Jun;12(3):174-179. doi: 10.1097/IMI.0000000000000376. PMID 28549028
- [Background] Harskamp RE, Puskas JD, Tijssen JG, Walker PF, Liberman HA, Lopes RD, Vassiliades TA, Peterson ED, Halkos ME. Comparison of hybrid coronary revascularization versus coronary artery bypass grafting in patients>/=65 years with multivessel coronary artery disease. Am J Cardiol. 2014 Jul 15;114(2):224-9. doi: 10.1016/j.amjcard.2014.04.028. Epub 2014 May 2. PMID 24878119
- [Background] Harskamp RE, Bagai A, Halkos ME, Rao SV, Bachinsky WB, Patel MR, de Winter RJ, Peterson ED, Alexander JH, Lopes RD. Clinical outcomes after hybrid coronary revascularization versus coronary artery bypass surgery: a meta-analysis of 1,190 patients. Am Heart J. 2014 Apr;167(4):585-92. doi: 10.1016/j.ahj.2014.01.006. Epub 2014 Jan 29. PMID 24655709
- [Background] Lowenstern A, Wu J, Bradley SM, Fanaroff AC, Tcheng JE, Wang TY. Current landscape of hybrid revascularization: A report from the NCDR CathPCI Registry. Am Heart J. 2019 Sep;215:167-177. doi: 10.1016/j.ahj.2019.06.014. Epub 2019 Jun 28. PMID 31349108
- [Background] Gortzen Q, Sampon F, Timmermans N, Woorst JT, Akca F. Endoscopic-Assisted Multivessel Off-Pump Coronary Artery Bypass Grafting: Experience of the First 100 Procedures. J Chest Surg. 2025 Jan 5;58(1):21-30. doi: 10.5090/jcs.24.080. Epub 2024 Nov 18. PMID 39552038
- [Background] Sampon F, Ter Woorst J, Dekker L, Akca F. Thoracoscopic-assisted, minimally invasive versus off-pump bypass grafting for single vessel coronary artery disease - A propensity matched analysis. Int J Cardiol. 2024 Aug 15;409:132175. doi: 10.1016/j.ijcard.2024.132175. Epub 2024 May 14. PMID 38754586
- [Background] Akca F. Thoracoscopic (non-robotic) harvesting of bilateral internal mammary artery grafts. Multimed Man Cardiothorac Surg. 2023 Nov 15;2023. doi: 10.1510/mmcts.2023.069. PMID 37965985
- [Background] Chen S, Karmpaliotis D, Redfors B, Shlofmitz E, Ben-Yehuda O, Crowley A, Mehdipoor G, Puskas JD, Kandzari DE, Banning AP, Morice MC, Taggart DP, Sabik JF 3rd, Serruys PW, Kappetein AP, Stone GW. Does an occluded RCA affect prognosis in patients undergoing PCI or CABG for left main coronary artery disease? Analysis from the EXCEL trial. EuroIntervention. 2019 Aug 9;15(6):e531-e538. doi: 10.4244/EIJ-D-19-00263. PMID 31186220
- [Background] Sajja LR, Mannam G. Internal thoracic artery: anatomical and biological characteristics revisited. Asian Cardiovasc Thorac Ann. 2015 Jan;23(1):88-99. doi: 10.1177/0218492314523629. Epub 2014 Feb 11. PMID 24585304
- [Background] Royse AG, Brennan AP, Ou-Young J, Pawanis Z, Canty DJ, Royse CF. 21-Year Survival of Left Internal Mammary Artery-Radial Artery-Y Graft. J Am Coll Cardiol. 2018 Sep 18;72(12):1332-1340. doi: 10.1016/j.jacc.2018.06.064. PMID 30213324
- [Background] Head SJ, Milojevic M, Daemen J, Ahn JM, Boersma E, Christiansen EH, Domanski MJ, Farkouh ME, Flather M, Fuster V, Hlatky MA, Holm NR, Hueb WA, Kamalesh M, Kim YH, Makikallio T, Mohr FW, Papageorgiou G, Park SJ, Rodriguez AE, Sabik JF 3rd, Stables RH, Stone GW, Serruys PW, Kappetein AP. Mortality after coronary artery bypass grafting versus percutaneous coronary intervention with stenting for coronary artery disease: a pooled analysis of individual patient data. Lancet. 2018 Mar 10;391(10124):939-948. doi: 10.1016/S0140-6736(18)30423-9. Epub 2018 Feb 23. PMID 29478841
- [Background] Fearon WF, Zimmermann FM, De Bruyne B, Piroth Z, van Straten AHM, Szekely L, Davidavicius G, Kalinauskas G, Mansour S, Kharbanda R, Ostlund-Papadogeorgos N, Aminian A, Oldroyd KG, Al-Attar N, Jagic N, Dambrink JE, Kala P, Angeras O, MacCarthy P, Wendler O, Casselman F, Witt N, Mavromatis K, Miner SES, Sarma J, Engstrom T, Christiansen EH, Tonino PAL, Reardon MJ, Lu D, Ding VY, Kobayashi Y, Hlatky MA, Mahaffey KW, Desai M, Woo YJ, Yeung AC, Pijls NHJ; FAME 3 Investigators. Fractional Flow Reserve-Guided PCI as Compared with Coronary Bypass Surgery. N Engl J Med. 2022 Jan 13;386(2):128-137. doi: 10.1056/NEJMoa2112299. Epub 2021 Nov 4. PMID 34735046
- [Background] Holm NR, Makikallio T, Lindsay MM, Spence MS, Erglis A, Menown IBA, Trovik T, Kellerth T, Kalinauskas G, Mogensen LJH, Nielsen PH, Niemela M, Lassen JF, Oldroyd K, Berg G, Stradins P, Walsh SJ, Graham ANJ, Endresen PC, Frobert O, Trivedi U, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in the treatment of unprotected left main stenosis: updated 5-year outcomes from the randomised, non-inferiority NOBLE trial. Lancet. 2020 Jan 18;395(10219):191-199. doi: 10.1016/S0140-6736(19)32972-1. Epub 2019 Dec 23. PMID 31879028
- [Background] Farkouh ME, Domanski M, Sleeper LA, Siami FS, Dangas G, Mack M, Yang M, Cohen DJ, Rosenberg Y, Solomon SD, Desai AS, Gersh BJ, Magnuson EA, Lansky A, Boineau R, Weinberger J, Ramanathan K, Sousa JE, Rankin J, Bhargava B, Buse J, Hueb W, Smith CR, Muratov V, Bansilal S, King S 3rd, Bertrand M, Fuster V; FREEDOM Trial Investigators. Strategies for multivessel revascularization in patients with diabetes. N Engl J Med. 2012 Dec 20;367(25):2375-84. doi: 10.1056/NEJMoa1211585. Epub 2012 Nov 4. PMID 23121323
- [Background] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612
- [Background] Virani SS, Newby LK, Arnold SV, Bittner V, Brewer LC, Demeter SH, Dixon DL, Fearon WF, Hess B, Johnson HM, Kazi DS, Kolte D, Kumbhani DJ, LoFaso J, Mahtta D, Mark DB, Minissian M, Navar AM, Patel AR, Piano MR, Rodriguez F, Talbot AW, Taqueti VR, Thomas RJ, van Diepen S, Wiggins B, Williams MS; Peer Review Committee Members. 2023 AHA/ACC/ACCP/ASPC/NLA/PCNA Guideline for the Management of Patients With Chronic Coronary Disease: A Report of the American Heart Association/American College of Cardiology Joint Committee on Clinical Practice Guidelines. Circulation. 2023 Aug 29;148(9):e9-e119. doi: 10.1161/CIR.0000000000001168. Epub 2023 Jul 20. PMID 37471501
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] World Health Organization. The top 10 causes of death. Published August 7, 2024. Accessed July 16, 2025. https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death
- [Background] Gortzen Q, Sampon F, Timmermans N, Ter Woorst J, Akca F. Endoscopic-assisted, minimally invasive versus sternotomy total arterial multivessel bypass grafting. Interdiscip Cardiovasc Thorac Surg. 2024 Nov 6;39(5):ivae187. doi: 10.1093/icvts/ivae187. PMID 39540774